CLINICAL TRIAL: NCT04648943
Title: The Effect of Antiglaucoma Procedures (Trabeculectomy vs. Ex-PRESS Glaucoma Drainage Implant) on the Corneal Biomechanical Properties
Brief Title: The Effect of Trabeculectomy & Ex-PRESS Glaucoma Drainage Implant on the Corneal Biomechanical Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES8/Th11/10-10-2013
Record Dates: First submitted 2020-11-21; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Glaucoma Eye
Keywords: glaucoma; trabeculectomy; Ex-PRESS glaucoma drainage implant; corneal hysteresis; corneal resistance factor
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing Ex-Press mini shunt insertion (Active Comparator): Patients in this arm had the Ex-Press mini shunt inserted in the operated eye in order to reduce the Intraocular Pressure. The corneal biomechanical properties were measured before and at 1, 6 and 12 months after surgery with the Ocular Response Analyzer
  Interventions: Procedure: Ex-Press mini shunt insertion
- Patients undergoing trabeculectomy (Active Comparator): Patients in this arm had standard trabeculectomy in the operated eye in order to reduce the Intraocular Pressure. The corneal biomechanical properties were measured before and at 1, 6 and 12 months after surgery with the Ocular Response Analyzer
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Procedure: Ex-Press mini shunt insertion
  Arms: Patients undergoing Ex-Press mini shunt insertion
Procedure: Trabeculectomy
  Arms: Patients undergoing trabeculectomy

SUMMARY:
This study aims to look into the change of the corneal biomechanical properties in patients undergoing insertion of the Ex-PRESS mini shunt or trabeculectomy for medically uncontrolled glaucoma

DETAILED DESCRIPTION:
The patients in the study were divided into two groups. In group 1 the patients had the Ex-PRESS mini shunt inserted in the operated eye and in group 2 the patients underwent standard trabeculectomy.

The corneal biomechanical properties were measured with the Ocular Response Analyzer before surgery and at 1, 6 and 12 months after surgery. The corneal biomechanical properties measured were the Corneal Hysteresis (CH) and the Corneal Resistance Factor (CRF).

The change of the CH and CRF was compared in each group before and after surgery (at the aforementioned predetermined time points) and between the two groups.

The intraocular pressure was also measured with the Goldmann applanation tonometer at the same time points and the change was compared before and after surgery in each group and between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Average Intraocular pressure > 24 mmHg on at least 2 occasions 1 month before surgery
* Congenital glaucoma

Exclusion Criteria:

* Previous ocular trauma
* Previous ocular surgery other than phacoemulsification
* Previous disease of the ocular surface

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change of corneal biomechanical properties | 12 months
  Two corneal biomechanical properties were measured with the use of the Ocular Response Analyzer (ORA): the Corneal Resistance Factor (CRF) and the Corneal Hysteresis (CH).
  These two indicators were measured before surgery and at 1, 6 and 12 months after surgery

SECONDARY OUTCOMES:
Change of Intraocular Pressure | 12 months
  The Intraocular Pressure was measured with the Goldmann applanation tonometer before surgery and at 1, 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece